CLINICAL TRIAL: NCT04229355
Title: Drug-eluting Bead Transarterial Chemoembolization Plus Lenvatinib or Sorafenib or PD-1 Inhibitor for Unresectable Hepatocellular Carcinoma: a Multicentric Prospective Study
Brief Title: DEB-TACE Plus Lenvatinib or Sorafenib or PD-1 Inhibitor for Unresectable Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Jian-Hong Zhong, Professor, Guangxi Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DEEP
Record Dates: First submitted 2020-01-12; First posted 2020-01-18 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib; lenvatinib; Immune Checkpoint Inhibitors

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will be blinded about patients' allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DEB-TACE plus Sorafenib (Experimental): Patients with unresectable hepatocellular carcinoma (HCC) in this group will receive drug-eluting bead transarterial chemoembolization (DEB-TACE).And then, they will receive sorafenib (400 mg/d, po, bid) one week after DEB-TACE therapy. The second DEB-TACE will be performed after one month later the first DEB-TACE. Lenvatinib will be taken orally for six months, untill tumor progression, or intolerable adverse reactions.
  Interventions: Drug: DEB-TACE plus Sorafenib
- DEB-TACE plus Lenvatinib (Experimental): Patients with unresectable hepatocellular carcinoma (HCC) in this group will receive drug-eluting bead transarterial chemoembolization (DEB-TACE).And then, they will receive lenvatinib (8 mg/d, po, qd) one week after DEB-TACE therapy. The second DEB-TACE will be performed after one month later the first DEB-TACE. Lenvatinib will be taken orally for six months, untill tumor progression, or intolerable adverse reactions.
  Interventions: Drug: DEB-TACE plus Lenvatinib
- DEB-TACE plus PD-1 inhibitor (Active Comparator): Patients with unresectable hepatocellular carcinoma (HCC) in this group will receive drug-eluting bead transarterial chemoembolization (DEB-TACE).And then, they will receive PD-1 inhibitor (200 mg, iv, 3 weeks) one week after DEB-TACE therapy. The second DEB-TACE will be performed after one month later the first DEB-TACE. PD-1 inhibitor will be taken for six months, untill tumor progression, or intolerable adverse reactions.
  Interventions: Drug: DEB-TACE plus PD-1 inhibitor

INTERVENTIONS:
Drug: DEB-TACE plus Sorafenib — Drug-eluting bead transarterial chemoembolization plus sorafenib (400 mg/d, po, bid)
  Arms: DEB-TACE plus Sorafenib
Drug: DEB-TACE plus Lenvatinib — Drug-eluting bead transarterial chemoembolization plus lenvatinib (8 mg/d, po, qd)
  Arms: DEB-TACE plus Lenvatinib
Drug: DEB-TACE plus PD-1 inhibitor — Drug-eluting bead transarterial chemoembolization plus PD-1 inhibitor
  Arms: DEB-TACE plus PD-1 inhibitor

SUMMARY:
Transarterial chemoembolization (TACE) based on drug-eluting beads (DEB-TACE) is widely used for unresectable hepatocellular carcinoma (HCC). However, the long-term survival is still low after DEB-TACE treatment. In recent years, lenvatinib and anti-PD-1 have exhibited potential therapeutic effects for advanced HCC. And sorafenib is the standard drug for advanced HCC. Combining targeted drugs or immunotherapies with DEB-TACE may provide synergistic effects and facilitate the development of personalized medicine. Therefore, this prospective study aims to investigate the safety and efficacy of DEB-TACE plus sorafenib or lenvatinib or PD-1 Inhibitor for unresectable HCC.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the most common type of liver cancer. Most patients with HCC are diagnosed as advanced stage or unresectable disease because of the lack of signs and symptoms. Despite significant research efforts, only a few effective treatment approaches have been developed for HCC. Conventional transarterial chemoembolization (cTACE) is widely used as a palliative treatment for inoperable HCC. TACE based on drug-eluting beads (DEB-TACE) has recently been introduced into the clinic. This technique relies on drug-loaded microspheres to embolize and release antitumor medication gradually and locally in order to maximize local ischemia and tumor necrosis. Nowadays, many RCTs and meta-analyses found DEB-TACE is associated with higher overall survival than cTACE for unresectable HCC. However, the long-term survival is still low after DEB-TACE treatment. In recent years, targeted drugs (such as sorafenib, lenvatinib) and immune checkpoint inhibitor (anti-PD-1) have exhibited potential therapeutic effects for advanced HCC. Lenvatinib is non-inferior to sorafenib in overall survival in untreated advanced HCC. Combining targeted drugs or immunotherapies with conventional therapeutic approaches may provide synergistic effects and facilitate the development of personalized medicine. However, it is still unknown which is the best combining treatment. Therefore, this prospective study aims to investigate the safety and efficacy of DEB-TACE plus sorafenib or lenvatinib or PD-1 Inhibitor for unresectable HCC.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 75 years
* Patients with unresectable primary hepatocellular carcinoma.
* With Child-Pugh A liver function.

Exclusion Criteria:

* Patients received targeted drugs, anti-PD1, or anti-PD-L1 treatment.
* Patients with recurrent hepatocellular carcinoma.
* Patient compliance is poor.
* The blood supply of tumor lesions is absolutely poor or arterial-venous shunt that TACE can not be performed.
* Known history of human immunodeficiency virus (HIV) infection.
* Known Central Nervous System tumors including metastatic brain disease.
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* History of organ allograft.
* Known or suspected allergy to the investigational agent or any agent given in association with this trial.
* Any condition that is unstable or which could jeopardize the safety of the patient and his/her compliance in the study.
* Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed within seven days prior to the start of study drug. Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-02-02 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | one month
  Primary endpoint is progression-free survival (PFS).

SECONDARY OUTCOMES:
Overall survival | one month
  Overall survival is measured from the date of enrollment until the date of death from any cause. Patients who is lost to follow-up are censored at the last date they are known to be alive, and patients who remain alive are censored at the time of data cutoff.

CONTACTS AND LOCATIONS:
Overall Officials: Le-Qun Li, PhD, Study Chair — Guangxi Medical University Cancer Hospital
Locations (1):
- Guangxi Medical University Cancer Hospital, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kudo M, Finn RS, Qin S, Han KH, Ikeda K, Piscaglia F, Baron A, Park JW, Han G, Jassem J, Blanc JF, Vogel A, Komov D, Evans TRJ, Lopez C, Dutcus C, Guo M, Saito K, Kraljevic S, Tamai T, Ren M, Cheng AL. Lenvatinib versus sorafenib in first-line treatment of patients with unresectable hepatocellular carcinoma: a randomised phase 3 non-inferiority trial. Lancet. 2018 Mar 24;391(10126):1163-1173. doi: 10.1016/S0140-6736(18)30207-1. PMID 29433850
- [Background] Hatanaka T, Kakizaki S, Nagashima T, Namikawa M, Tojima H, Shimada Y, Takizawa D, Naganuma A, Arai H, Sato K, Harimoto N, Shirabe K, Uraoka T. Analyses of objective response rate, progression-free survival, and adverse events in hepatocellular carcinoma patients treated with lenvatinib: A multicenter retrospective study. Hepatol Res. 2020 Mar;50(3):382-395. doi: 10.1111/hepr.13460. Epub 2019 Dec 10. PMID 31760660
- [Background] Kim JJ, McFarlane T, Tully S, Wong WWL. Lenvatinib Versus Sorafenib as First-Line Treatment of Unresectable Hepatocellular Carcinoma: A Cost-Utility Analysis. Oncologist. 2019 Nov 20:theoncologist.2019-0501. doi: 10.1634/theoncologist.2019-0501. Online ahead of print. PMID 31748341
- [Background] Feng Z, Rong P, Wang W. Meta-analysis of the efficacy and safety of PD-1/PD-L1 inhibitors administered alone or in combination with anti-VEGF agents in advanced hepatocellular carcinoma. Gut. 2020 Oct;69(10):1904-1906. doi: 10.1136/gutjnl-2019-320116. Epub 2019 Dec 18. No abstract available. PMID 31852768
- [Background] Xie ZB, Wang XB, Peng YC, Zhu SL, Ma L, Xiang BD, Gong WF, Chen J, You XM, Jiang JH, Li LQ, Zhong JH. Systematic review comparing the safety and efficacy of conventional and drug-eluting bead transarterial chemoembolization for inoperable hepatocellular carcinoma. Hepatol Res. 2015 Jan;45(2):190-200. doi: 10.1111/hepr.12450. Epub 2014 Dec 24. PMID 25388603